CLINICAL TRIAL: NCT02857010
Title: Therapeutic Effects of Allogenic Mesenchymal Stem Cells in Cirrhotic Patients With Acute-on-chronic Liver Failure. A Double-blind Randomized Placebo-controlled Trial
Brief Title: Allogenic Bone Marrow Mesenchymal Stem Cell Therapy in Acute-on-chronic Liver Failure
Acronym: Liveradvance
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Dificulties to recruit patients and dificulties to obtain MSCs.
Sponsor: Pere Gines (Other)
Collaborators: Clinica Universidad de Navarra, Universidad de Navarra (Other)
Responsible Party: Sponsor-Investigator, Pere Gines, Head of the Liver Unit, Hospital Clinic of Barcelona
Organization: Hospital Clinic of Barcelona (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2012-003900-11
Record Dates: First submitted 2016-03-08; First posted 2016-08-05 (Estimated); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Acute on Chronic Hepatic Failure

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Allogenic Mesenchymal stem cells (Experimental): Intravenous allogenic bone marrow derived mesenchymal stem cells: 4 doses of 2 x 106/kg administered on days 1, 4, 11 and 18
  Interventions: Biological: Allogenic mesenchymal stem cells
- Placebo (Placebo Comparator): Solution without cells on days 1, 4, 11 and 18
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Allogenic mesenchymal stem cells — Cell therapy
  Arms: Allogenic Mesenchymal stem cells
Other: Placebo — Serum without stem cells
  Arms: Placebo

SUMMARY:
Double-blind placebo randomized controlled trial evaluating the clinical efficacy of allogenic bone marrow derived mesenchymal stem cells in cirrhotic patients with acute-on-chronic liver failure

DETAILED DESCRIPTION:
Introduction: The most important cause of death in patients with cirrhosis is the development of Acute-on-Chronic Liver Failure (ACLF), a syndrome recently redefined with high mortality. The only effective treatment for ACLF is liver transplantation. However, available organs are limited. Other treatments, such as artificial liver support systems, do not improve survival. ACLF is characterized by increased systemic inflammatory state together with impaired liver regeneration what leads to multiorgan failure. Mesenchymal stem cell (MSC) therapy is an attractive strategy for ACLF owing to the immunomodulatory and regenerative properties of these cells. Aim: To investigate the effects of allogeneic bone marrow MSCs transplantation on liver and other organ functions and systemic inflammation in patients with ACLF. Altruist bone marrow donors will be the source of MSCs. Design and methodology: randomized, double-blind phase I placebo-controlled trial aimed at comparing placebo (solution without cells) and MSCs (4 doses of 2 x 106/kg administered on days 1, 4, 11 and 18). Thirty patients, 15 per group will be included. ACLF will be defined by the CLIF SOFA score and patients stratified according to severity. Outcomes evaluated will be: 1) Organ function (CLIF SOFA and CLIF-C ACLF score); 2) Liver (Child-Pugh and MELD scores,serum bile acids, ammonia and lactate levels), circulatory (systemic and splanchnic hemodynamics, renin, noradrenalin) and endothelial function (nitric oxide, von Willebrand factor); 3 Inflammatory response (serum cytokine panel and transcriptomic analysis of monocytes and polymorphonuclear cells from peripheral blood); 4) Survival at 28 days, 3 and 12 months; and 5) Safety. Expected results: Therapy with MSCs could have beneficial effects on the evolution of patients with ACLF (modulation of inflammatory response and improvement of liver and extra-hepatic organ function) what could translate into an improvement on short-term survival.

ELIGIBILITY:
Inclusion Criteria:

* Liver cirrhosis
* ACLF grade 1, 2 or 3 (Canonic criteria)
* Signed informed consent

Exclusion Criteria:

* Acute or subacute liver failure without cirrhosis
* ACLF grade 1 with response to medical therapy
* Evidence of current malignancy including hepatocellular carcinoma (any grade) or alphafetoprotein > 400 ng/ml
* Previous personal history of malignancy (active or in complete remission) or familiar history of hereditary cancer.
* Moderate or severe chronic heart failure (NYHA III-IV)
* Renal replacement therapy
* Severe chronic pulmonary disease (GOLD III-IV)
* Gastrointestinal bleeding in the last 5 days
* Previous liver transplantation
* Immunosuppressive therapy
* Extrahepatic cholestasis
* HIV infection
* Pregnant of breastfeeding women
* Pre-menopausal women who are of child bearing potential and are not practicing an acceptable method of birth control.
* Participation in any investigational trial in the last 3 months
* Active addition to illegal drugs
* Refusal to participate
* Patients who can not provide prior informed consent

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2020-02 (Actual)

PRIMARY OUTCOMES:
Change in organ function: chronic liver failure-sequential organ failure assessment (CLIF-SOFA) | Change from Baseline CLIF-SOFA score at 28 days

SECONDARY OUTCOMES:
Child-Pugh score as a marker of liver function | Change from Baseline Child-Pugh score at 28 days, 90 days, one year and 2 years
  Child-Pugh
Model for End-stage Liver Disease (MELD) score as a marker of liver function | Change from Baseline MELD score at 28 days, 90 days, one year and 2 years
  MELD scores
serum bile acids as a surrogate marker of liver function | Change from Baseline serum bile acids at 28 days
  serum bile acids
ammonia levels as a surrogate marker of liver function | Change from Baseline serum ammonia at 7, 21 and 28 days
  ammonia
Lactate levels as a surrogate marker of liver function | Change from Baseline serum lactate levels at 7, 21 and 28 days
  lactate levels
Hepatic portal venous gradient (HPVG) | Change from Baseline HPVG at 21 days
  HPVG in mmHg
Endothelial function measured by nitric oxide levels | Change from Baseline serum nitric oxide levels at 7, 21 and 28 days
  Nitric oxide
Endothelial function measured by von Willebrand factor levels | Change from Baseline serum von Willebrand factor levels at 7, 21 and 28 days
  von Willebrand factor
Renal function measured by serum creatinine | Change from Baseline serum creatinine at 7, 21 and 28 days
  serum creatinine
Renal function measured by Blood urea nitrogen (BUN) | Change from Baseline serum BUN at 7, 21 and 28 days
  serum BUN
urine neutrophil gelatinase-associated lipocalin (NGAL) as a surrogate marker of renal function | Change from Baseline NGAL at 7, 21 and 28 days
  urine neutrophil gelatinase-associated lipocalin (NGAL)
Inflammatory response | Change from Baseline cytokine panel at 4, 11 and 18 days
  Serum cytokine panel
Transcriptome analysis | Change from Baseline transcriptome analysis at 7-8 days and 12-18 days
  Transcriptome analysis of monocytes and polymorphonuclear cells from peripheral blood
Number of participants alive | Number of participants alive at 28 days, 3 months, 12 months and 2 years
Number of participants with treatment-related adverse events as assessed by World Health Organization (WHO) classification for acute and subacute toxicity | Number of participants with treatment-related adverse events as assessed by WHO classification for acute and subacute toxicity at 2 years
Change in chronic liver failure C acute on chronic liver failure score (clif C ACLF) | Change from Baseline clif C ACLF score at 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Javier Fernandez, MD, PhD, Study Chair — Hospital Clinic
Locations (1):
- Hospital Clinic de Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes